CLINICAL TRIAL: NCT01493310
Title: A Randomized Phase I Trial of Nanoparticle Albumin Bound Paclitaxel (Nab-paclitaxel, Abraxane) With or Without Mifepristone for Advanced Breast Cancer
Brief Title: Nab-paclitaxel (Abraxane) With or Without Mifepristone in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0546; NCI-2011-03525 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-02; First posted 2011-12-15 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Mifepristone; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (hormone therapy, chemotherapy) (Experimental): Patients will receive mifepristone and nab-paclitaxel in 28-day treatment cycles. Patients receive mifepristone once a day by mouth on days 0, 1, 7, 8, 14, and 15 and nab-paclitaxel by intravenous infusion (IV) on days 1, 8, and 15. Treatment cycles are repeated every 28 days in the absence of disease progression or unacceptable side effects.
  Interventions: Drug: mifepristone; Drug: nab-paclitaxel
- Arm B (chemotherapy) (Active Comparator): Patients will receive nab-paclitaxel and placebo for a 28-day treatment cycle (Cycle 1).
  Patients receive placebo once a day by mouth on days 0, 1, 7, 8, 14, and 15 and nab-paclitaxel by intravenous infusion (IV) on days 1, 8, and 15. Patients then cross-over to Arm A after completion of the first treatment cycle.
  Interventions: Drug: placebo; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: mifepristone — Given orally (by mouth)
  Up to 4 doses of mifepristone will be studied (300 mg, 600 mg, 900 mg, 1200 mg)
  Other Names: Mifegyne; Mifeprex; RU-38486
  Arms: Arm A (hormone therapy, chemotherapy)
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm B (chemotherapy)
Drug: nab-paclitaxel — Given by intravenous infusion (IV)
  Dose of 80 mg/m2
  Other Names: ABI-007; nab paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; nanoparticle albumin-bound paclitaxel

SUMMARY:
This trial will find the best dose of mifepristone when given together with nab-paclitaxel (Abraxane) based on the side effects of the two drugs in patients with advanced breast cancer.

Patients will be randomized to receive nab-paclitaxel with or without mifepristone during the first treatment cycle. After the first cycle, all patients will receive nab-paclitaxel with mifepristone until their disease worsens or they experience an unacceptable side effect.

This study will test up to 4 doses of mifepristone in combination with nab-paclitaxel. The study will first test the lowest dose in a small group of patients and if they do not have bad side effects, higher doses will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic (stage IV) or unresectable (cannot be removed by surgery) stage III breast cancer
* Patients must have evaluable disease
* Patients may have received adjuvant chemotherapy and up to four prior chemotherapy regimens for metastatic or locally recurrent disease and cannot have received prior nab-paclitaxel or mifepristone therapy for metastatic disease
* Patients who are estrogen receptor (ER)- and/or progesterone receptor (PR)-positive must have developed metastatic disease while on adjuvant hormonal therapy or have progression of disease after at least one hormonal therapy for advanced disease) and may have received unlimited prior hormonal therapies
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky > 60%)
* Absolute neutrophil count >= 1,500/mL
* Platelets >= 100,000/mL
* Total bilirubin =< institutional upper limit of normal (ULN)
* AST (serum glutamic oxaloacetic transaminase [SGOT])/ALT (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN
* Creatinine =< institutional ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Morning cortisol >= institutional normal
* Negative serum or urine pregnancy test is required for women of child-bearing potential (able to get pregnant)
* Women of child-bearing potential and men who are sexually active must agree to use two forms of birth control prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational drugs or treatments
* Patients with known brain metastases are eligible as long as they have completed radiation to the brain and have been off of corticosteroid therapy for at least 4 weeks
* History of allergic reactions to compounds similar to mifepristone or paclitaxel/nab-paclitaxel; patients with a history of mild infusion reactions with paclitaxel who were able to continue to receive paclitaxel with corticosteroid premedications will be eligible to participate, as these cases were likely related to Cremophor and not paclitaxel
* Mifepristone may affect the way the body processes some types of drugs so they cannot be taken while on-study. These include but are not limited to non-steroidal anti-inflammatory drugs (NSAIDs) or warfarin, cyclosporine, certain benzodiazepines. The study doctor will review patient's current medications to determined if any are prohibited from the study.
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if patient wishes to participate in the study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* No history of long-term or ongoing short term use of corticosteroids is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Determination of the safest dose of mifepristone when given in combination with nab-paclitaxel | 28days (Cycle 1)
  This study will seek the safest dose of mifepristone given in combination with nab-paclitaxel. Safety of each dose will be determined by the number and seriousness of side effects experienced by patients receiving each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nanda, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois